CLINICAL TRIAL: NCT01877265
Title: Assessment of the Impact of Monomethoxy Polyethylene Glycols on the Pharmacokinetics and Glucodynamics of Single Doses of LY2605541 in Healthy Subjects
Brief Title: A Study of LY2605541 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 14594; I2R-MC-BIDH (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — LY2605541

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY2605541 - Source 1 (Experimental): Each healthy participant will receive a single subcutaneous (SC) injection of 0.5 units per kilogram (U/kg) of LY2605541 on Day 1 of 1 of 3 treatment periods
  Interventions: Drug: LY2605541
- LY2605541 - Source 2 (Experimental): Each healthy participant will receive single SC injection of 0.5 U/kg of LY2605541 on Day 1 of 1of 3 treatment periods
  Interventions: Drug: LY2605541
- LY2605541 - Source 3 (Experimental): Each healthy participant will receive single SC injection of 0.5 U/kg of LY2605541 on Day 1 of 1 of 3 treatment periods
  Interventions: Drug: LY2605541

INTERVENTIONS:
Drug: LY2605541

SUMMARY:
This study looks at the amount of LY2605541 in the body after it is injected under the skin. The study has 3 periods, each lasting 10 days. Each participant will receive one injection in each period. At least 14 days will pass between each injection.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* A body mass index of 18.5 to 30 kilograms per meter square (kg/m^2)

Exclusion Criteria:

* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Are women with a positive pregnancy test or are women who are lactating
* Intend to use over-the-counter medication within 7 days prior to dosing or prescription medication within 14 days prior to dosing (apart from contraceptive medication, vitamin/mineral supplements, occasional acetaminophen, and/or hormone replacement therapy)
* Have donated blood of more than 500 milliliters (mL) within the last month
* Have an average weekly alcohol intake that exceeds 21 units per week (for males) and 14 units per week (for females)
* Are excessive consumers of xanthines (more than 10 cups of tea, coffee, cola, or hot chocolate per day)
* Have a fasting blood glucose (BG) >110 milligrams per deciliter (mg/dL) (6.1 millimoles per liter [mmol/L])
* Currently smoke more than 10 cigarettes per day, or are unwilling to refrain from smoking for 72 hours prior to each dosing occasion and during confinement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: LY2605541 was manufactured using the 3 different polyethylene glycol (PEG) sources (referred to as Source 1 [LY1], Source 2 [LY2], and Source 3 [LY3]). Participants were randomized to 1 of 6 treatment sequences and received a single injection of LY1, LY2, or LY3 on Day 1 of each of 3 treatment periods according to their assigned treatment sequence.
Groups:
- LY3/LY2/LY1: A single, subcutaneous (SC) injection of 0.5 units per kilogram (U/kg) LY2605541 from Source 3 on Day 1 of Period 1; from Source 2 on Day 1 of Period 2; and from Source 1 on Day 1 of Period 3.
  There was a washout period of at least 14 days between injections. Each participant received up to 3 injections.
- LY2/LY1/LY3: A single, SC injection of 0.5 U/kg LY2605541 from Source 2 on Day 1 of Period 1; from Source 1 on Day 1 of Period 2; and from Source 3 on Day 1 of Period 3.
  There was a washout period of at least 14 days between injections. Each participant received up to 3 injections.
- LY1/LY2/LY3: A single, SC injection of 0.5 U/kg LY2605541 from Source 1 on Day 1 of Period 1; from Source 2 on Day 1 of Period 2; and from Source 3 on Day 1 of Period 3.
  There was a washout period of at least 14 days between injections. Each participant received up to 3 injections.
- LY1/LY3/LY2: A single, SC injection of 0.5 U/kg LY2605541 from Source 1 on Day 1 of Period 1; from Source 3 on Day 1 of Period 2; and from Source 2 on Day 1 of Period 3.
  There was a washout period of at least 14 days between injections. Each participant received up to 3 injections.
- LY3/LY1/LY2: A single, SC injection of 0.5 U/kg LY2605541 from Source 3 on Day 1 of Period 1; from Source 1 on Day 1 of Period 2; and from Source 2 on Day 1 of Period 3.
  There was a washout period of at least 14 days between injections. Each participant received up to 3 injections.
- LY2/LY3/LY1: A single, SC injection of 0.5 U/kg LY2605541 from Source 2 on Day 1 of Period 1; from Source 3 on Day 1 of Period 2; and from Source 1 on Day 1 of Period 3.
  There was a washout period of at least 14 days between injections. Each participant received up to 3 injections.
Period: Treatment Period 1
Arm/Group | LY3/LY2/LY1 | LY2/LY1/LY3 | LY1/LY2/LY3 | LY1/LY3/LY2 | LY3/LY1/LY2 | LY2/LY3/LY1
Started | 3 | 3 | 3 | 3 | 3 | 3
Received at Least One Dose of Study Drug | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 1 | 0 | 0 | 0
Period: Washout Period 1 (at Least 14 Days)
Arm/Group | LY3/LY2/LY1 | LY2/LY1/LY3 | LY1/LY2/LY3 | LY1/LY3/LY2 | LY3/LY1/LY2 | LY2/LY3/LY1
Started | 3 | 3 | 2 | 3 | 3 | 3
Completed | 3 | 3 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | LY3/LY2/LY1 | LY2/LY1/LY3 | LY1/LY2/LY3 | LY1/LY3/LY2 | LY3/LY1/LY2 | LY2/LY3/LY1
Started | 3 | 3 | 2 | 3 | 3 | 3
Received at Least One Dose of Study Drug | 3 | 3 | 2 | 3 | 3 | 3
Completed | 3 | 3 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (at Least 14 Days)
Arm/Group | LY3/LY2/LY1 | LY2/LY1/LY3 | LY1/LY2/LY3 | LY1/LY3/LY2 | LY3/LY1/LY2 | LY2/LY3/LY1
Started | 3 | 3 | 2 | 3 | 3 | 3
Completed | 3 | 3 | 2 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period 3
Arm/Group | LY3/LY2/LY1 | LY2/LY1/LY3 | LY1/LY2/LY3 | LY1/LY3/LY2 | LY3/LY1/LY2 | LY2/LY3/LY1
Started | 3 | 3 | 2 | 3 | 3 | 2
Received at Least One Dose of Study Drug | 3 | 3 | 2 | 3 | 3 | 2
Completed | 2 | 3 | 2 | 3 | 3 | 2
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of LY2605541.
Groups:
- 0.5 U/kg LY2605541: Participants randomized to receive a single, SC injection of 0.5 U/kg LY2605541 using 3 different PEG sources on Day 1 of each of 3 treatment periods, according to their assigned treatment sequence.
Arm/Group | 0.5 U/kg LY2605541
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Time Curve From Zero to Infinity (AUC[0-∞]) of LY2605541
Description: LY2605541 exposure in terms of AUC from time 0 extrapolated to infinity (AUC[0-inf]) is summarized for each PEG source (LY1, LY2, or LY3).
Time Frame: Predose and 2, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, and 216 hours post dose in each period
Population: Participants who received at least 1 dose of LY2605541 and had evaluable LY2605541 concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles times hours per liter
Groups:
- 0.5 U/kg LY2605541 (LY1): LY2605541: 0.5 U/kg SC injection, single dose from PEG source 1 (LY1) on Day 1 of 1 of the 3 treatment periods.
- 0.5 U/kg LY2605541 (LY2): LY2605541: 0.5 U/kg SC injection, single dose from PEG source 2 (LY2) on Day 1 of 1 of the 3 treatment periods.
- 0.5 U/kg LY2605541 (LY3): LY2605541: 0.5 U/kg SC injection, single dose from PEG source 3 (LY3) on Day 1 of 1 of the 3 treatment periods.
Arm/Group | 0.5 U/kg LY2605541 (LY1) | 0.5 U/kg LY2605541 (LY2) | 0.5 U/kg LY2605541 (LY3)
Number analyzed (Participants) | 17 | 17 | 17
picomoles times hours per liter | 128000 (23) | 145000 (22) | 135000 (18)

2. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY2605541
Description: The maximum observed drug concentration (Cmax) of LY2605541 is summarized for each PEG source (LY1, LY2, or LY3).
Time Frame: Predose and 2, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, and 216 hours post dose in each period
Population: Participants who received at least 1 dose of LY2605541 and had evaluable LY2605541 concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles per liter
Groups:
- 0.5 U/kg LY2605541 (LY1): LY2605541: 0.5 U/kg SC injection, single dose from LY1 on Day 1 of 1 of the 3 treatment periods.
- 0.5 U/kg LY2605541 (LY2): LY2605541: 0.5 U/kg SC injection, single dose from LY2 on Day 1 of 1 of the 3 treatment periods.
- 0.5 U/kg LY2605541 (LY3): LY2605541: 0.5 U/kg SC injection, single dose from LY3 on Day 1 of 1 of the 3 treatment periods.
Arm/Group | 0.5 U/kg LY2605541 (LY1) | 0.5 U/kg LY2605541 (LY2) | 0.5 U/kg LY2605541 (LY3)
Number analyzed (Participants) | 17 | 17 | 17
picomoles per liter | 1980 (39) | 2490 (35) | 2210 (39)

3. Secondary Outcome: Glucodynamics: Maximum Glucose Infusion Rate (Rmax)
Description: The maximum observed glucose infusion rate following LY2605541 injection is summarized for each PEG source (LY1, LY2, or LY3).
Time Frame: Predose and up to 24 hours post dose in each period
Population: Participants who received at least 1 dose of LY2605541 and had evaluable glucose infusion data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per minute per kilogram
Arm/Group | 0.5 U/kg LY2605541 (LY1) | 0.5 U/kg LY2605541 (LY2) | 0.5 U/kg LY2605541 (LY3)
Number analyzed (Participants) | 17 | 17 | 17
milligrams per minute per kilogram | 1.21 (37) | 1.31 (57) | 1.40 (41)

4. Secondary Outcome: Glucodynamics: Total Amount of Glucose Infused (Gtot)
Description: The total amount of glucose infused following LY2605541 injection is summarized for each PEG source (LY1, LY2, or LY3).
Time Frame: Predose and up to 24 hours post dose in each period
Population: Participants who received at least 1 dose of LY2605541 and had evaluable glucose infusion data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per kilogram
Arm/Group | 0.5 U/kg LY2605541 (LY1) | 0.5 U/kg LY2605541 (LY2) | 0.5 U/kg LY2605541 (LY3)
Number analyzed (Participants) | 17 | 17 | 16
milligrams per kilogram | 900 (53) | 963 (103) | 1190 (49)

ADVERSE EVENTS:
Arm/Group | 0.5 U/kg LY2605541 (LY1) | 0.5 U/kg LY2605541 (LY2) | 0.5 U/kg LY2605541 (LY3)
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 4/17 | 6/17 | 3/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 U/kg LY2605541 (LY1) (N=17) | 0.5 U/kg LY2605541 (LY2) (N=17) | 0.5 U/kg LY2605541 (LY3) (N=17)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 2 (2) | 2 (2)
Catheter site swelling (General disorders) | 1 (2) | 1 (1) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days